CLINICAL TRIAL: NCT05473286
Title: A Multi-centre, Prospective, Non-interventional Single-arm Study Investigating Clinical Parameters Associated With the Use of Once-daily Oral Semaglutide in a Real-world Adult Population With Type 2 Diabetes in Germany
Brief Title: A Research Study Looking at How Oral Semaglutide Works in People With Type 2 Diabetes in Germany, as Part of Local Clinical Practice
Acronym: PIONEER REAL
Status: Withdrawn | Type: Observational
Why Stopped: Rybelsus® was not launched in Germany during the planned duration of NN9924-4540 study.
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN9924-4540
Record Dates: First submitted 2022-07-22; First posted 2022-07-25 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with type 2 diabetes: Adult patients with type 2 diabetes and naïve to injectable glucose-lowering treatment.
  Interventions: Drug: Oral Semaglutide

INTERVENTIONS:
Drug: Oral Semaglutide — Patients will be treated with commercially available oral semaglutide according to local label and to routine clinical practice at the discretion of the treating physician. The decision to initiate treatment with commercially available oral semaglutide has been made by the patient/Legally Acceptable Representative (LAR) and the treating physician based on local label before and independently from the decision to include the patient in this study.

SUMMARY:
The purpose of the study is to collect information on how Rybelsus® works in people with type 2 diabetes and to see if Rybelsus® can lower their blood sugar levels. Participants will get Rybelsus® as prescribed to them by the study doctor. The study will last for about 34-44 weeks. Participants will be asked to complete questionnaires about how they take their Rybelsus® tablets. Participants will complete the questionnaires during their normally scheduled visit with the study doctor.

ELIGIBILITY:
Inclusion Criteria:

* Signed consent obtained before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol).
* Diagnosed with type 2 diabetes mellitus.
* The decision to initiate treatment with commercially available oral semaglutide has been made by the patient/Legally Acceptable Representative (LAR) and the treating physician based on local label before and independently from the decision to include the patient in this study.
* Male or female, age above or equal to 18 years at the time of signing informed consent.
* Available HbA1c value less than or equal to (≤) 90 days prior to the 'Informed Consent and Treatment Initiation visit' (V1) or HbA1c measurement taken in relation with the 'Informed Consent and Treatment Initiation visit' (V1) if in line with local clinical practice.
* Treatment naïve to injectable glucose-lowering drug(s). An exception is short-term insulin treatment for acute illness for a total of less than (<) 14 days.

Exclusion Criteria:

* Previous participation in this study. Participation is defined as having given informed consent in this study.
* Treatment with any investigational drug within 30 days prior to enrolment into the study.
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients with type 2 diabetes and naïve to injectable glucose-lowering treatment.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-09-30 (Estimated); Primary Completion 2024-05-16 (Estimated); Study Completion 2024-05-16 (Estimated)

PRIMARY OUTCOMES:
Change in Glycated haemoglobin (HbA1c ) | From baseline (week 0) to End of Study visit (V3) (week 34-44)
  Percent-points.

SECONDARY OUTCOMES:
Relative change in body weight | From baseline (week 0) to End of Study visit (V3) (week 34-44)
  Percent.
Absolute change in body weight | From baseline (week 0) to End of Study visit (V3) (week 34-44)
  Kilogram (Kg).
HbA1c <7% (Yes or No) | End of Study visit (V3) (week 34-44)
  Percentage of patients achieving or not achieving HbA1c <7% (Yes or No).
HbA1c reduction >=1%-points and body weight reduction of >=5% (Yes/No) | From baseline (week 0) to End of Study visit (V3) (week 34-44)
  Percentage of patients achieving or not achieving HbA1c reduction >=1%-points and body weight reduction of >=5%.
HbA1c reduction >=1%-points and body weight reduction of >=3% (Yes/No) | From baseline (week 0) to End of Study visit (V3) (week 34-44)
  Percentage of patients achieving or not achieving HbA1c reduction >=1%-points and body weight reduction of >=3%.
Diabetes Treatment Satisfaction Questionnaire, change (DTSQc), relative treatment satisfaction | End of Study visit (V3) (week 34-44)
  The DTSQc provides a measure of how satisfied participants are with their current diabetes treatment compared with previous treatment. It consists of 8 questions, which are to be answered on a Likert scale from -3 to +3 (-3 = much less satisfied now to +3 = much more satisfied now), with 0 (midpoint), representing no change. Six questions are summed to produce a Total treatment satisfaction score. The remaining two questions concern perceived frequency of hyperglycemia and perceived frequency of hypoglycemia, respectively. The DTSQc Total treatment satisfaction score ranges from -18 to +18, with higher scores associated with greater treatment satisfaction.
Diabetes Treatment Satisfaction Questionnaire, status (DTSQs), change in absolute treatment satisfaction | From baseline (week 0) to End of Study visit (V3) (week 34-44)
  The DTSQs items are scored on a 7-point graded response scale ranging from 6 to 0. Higher scores indicate higher levels of treatment satisfaction for DTSQs items.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com